CLINICAL TRIAL: NCT03743129
Title: A Randomised, Open, Blank-controlled, Multi-centre Study of Anlotinib as Sequential Therapy in Patients With Unresectable NSCLC(Stage III) Who Have Not Progressed Following Definitive, Platinum-based, Concurrent Chemoradiation Therapy
Brief Title: Anlotinib After Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer（ALTER-L029）
Acronym: ALTER-L029
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Shi, MD (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Anhui Shi, MD, Associate Chief Physician, Peking University Cancer Hospital & Institute
Organization: Peking University Cancer Hospital & Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018YJZ47
Record Dates: First submitted 2018-11-11; First posted 2018-11-15 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Non-Small Cell Lung Cancer Stage III
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anlotinib (Experimental): Anlotinib p.o, qd. Treatment from Day 1 of randomization(after concurrent chemoradiation 4-6 weeks) to disease progress or untolerated toxicity or consent withdrawal. The 2:1 ratio (Anlotinib to blank).
  Interventions: Drug: Anlotinib
- Blank (No Intervention): No intervention from Day 1 of randomization(after concurrent chemoradiation 4-6 weeks) .The 2:1 ratio (Anlotinib to blank).

INTERVENTIONS:
Drug: Anlotinib — Anlotinib 12mg p.o, qd
  Other Names: AL3818
  Arms: Anlotinib

SUMMARY:
Evaluate the efficacy and safety of Anlotinib following concurrent chemoradiation in patients with stage III unresectable non-small cell lung cancer

DETAILED DESCRIPTION:
Anlotinib (AL3818) is a kind of innovative medicines approved by State Food and Drug Administration（SFDA:2011L00661） which was researched by Jiangsu Chia-tai Tianqing Pharmaceutical Co., Ltd. Anlotinib is a kinase inhibitor of receptor tyrosine with multi-targets, especially for VEGFR1、VEGFR2、VEGFR3、FGFR1/2/3、PDGFRa/β c-Kit and MET.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age at least 18 years.
* 2.Documented evidence of NSCLC (locally advanced, unresectable, Stage III).
* 3.Patients must have received at least 2 cycles of platinum-based chemotherapy concurrent with radiation therapy.
* 4.ECOG PS : 0 to 1.
* 5.Estimated life expectancy of more than 12 weeks.

Exclusion Criteria:

* 1.Prior exposure to any anti-angiogenesis drugs.
* 2.Central lung carcinoma along with large vessels or tumor with cavum or necrosis.
* 3.Evidence of severe or uncontrolled systemic diseases, including active bleeding diatheses or active infections including hepatitis B, C and HIV.
* 4.Any unresolved toxicity CTCAE >Grade 2 from the prior chemoradiation therapy.
* 5.Evidence of uncontrolled illness such as symptomatic congestive heart failure, uncontrolled hypertension or COPD.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Estimated to be from baseline up to 3 years
  the time from randomization until the date of objective disease progression (RECIST 1.1) or death (by any cause in the absence of progression)

SECONDARY OUTCOMES:
Disease Control Rate at 6 months(DCR6) | Estimated to be from baseline up to 3 years
  the percentage of patients with response of Complete Response (CR) or partial response (PR) or stable disease(SD) at least 4 weeks at 6 months after randomization
Disease Control Rate at 12 months(DCR12) | Estimated to be from baseline up to 3 years
  the percentage of patients with response of Complete Response (CR) or partial response (PR) or stable disease(SD) at least 4 weeks at 12 months after randomization
Overall Survival at 12 months (OS12) | Estimated to be from baseline up to 3 years
  the percentage of patients who are alive at 12 months after randomization per the Kaplan-Meier estimate of overall survival at 12 months
Overall Survival at 24 months (OS24) | Estimated to be from baseline up to 3 years
  the percentage of patients who are alive at 24 months after randomization per the Kaplan-Meier estimate of overall survival at 24 months
Recurrence rate at 12 months | Estimated to be from baseline up to 3 years
  the percentage of patients with Progressive Disease(PD) at 12 months after randomization
Recurrence rate at 24 months | Estimated to be from baseline up to 3 years
  the percentage of patients with Progressive Disease(PD) at 24 months after randomization

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The second hospital of Hebei Medical University, Shijiazhuang, Hebei

REFERENCES:
- [Derived] Yang D, Li X, Xue X, Jiang L, Shi A, Zhao J. Anlotinib hydrochloride consolidation after concurrent chemoradiotherapy in stage III non-small-cell lung cancer: a truncated, randomized, multicenter, clinical study (ALTER-L029). Anticancer Drugs. 2024 Aug 1;35(7):680-685. doi: 10.1097/CAD.0000000000001617. Epub 2024 May 3. PMID 38718190